CLINICAL TRIAL: NCT03923777
Title: Pilot Study Involving Active Surveillance With CT Imaging and Liquid BiOpsies iN Stage IA Lung Cancer (ACTION-Lung)
Brief Title: Active Surveillance in Early Lung Cancer
Acronym: ACTION-Lung
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Vermont Medical Center (Other)
Responsible Party: Principal Investigator, Christopher Anker, Radiation Oncology Physician, University of Vermont Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Chrms 18-0396
Record Dates: First submitted 2019-04-03; First posted 2019-04-23 (Actual); Last update posted 2020-07-16 (Actual); Status verified 2020-07

CONDITIONS: Stage IA Non-small Cell Lung Cancer; Lung Carcinoid Tumor
Keywords: Active Surveillance
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Watchful Waiting

STUDY DESIGN:
Intervention Model Description: Investigators propose a study involving active surveillance for NSCLC where patients would have consideration of SABR if either the tumor exceeded 3 cm in size or the volume doubling time (VDT) decreased to <400 days. Following enrollment, chest CT with contrast (with slice thickness ≤3 mm) to be performed 3 months (+/- 30 days) after the initial CT]. Patients with VDTs <400 days must be considered for SABR. SABR is not mandatory [patient choice] and active surveillance may be continued. Patients with VDTs ≥400 days continue active surveillance via serial CTs with intervals of every 3 months (+/- 30 days) up to 2 years total.
  Following informed consent, blood samples will be acquired following the protocol schedule based on enrollment group. Quality of life questionnaires will also be completed following the protocol schedule for the main cohort only.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Active Surveillance (Other): Active surveillance is a way of either delaying or avoiding treatment and its possible side effects through carefully watching for changes in the tumor. Patients continue on this regimen, watching for tumor growth, up to 2 years on study or until rate or extent of growth leads to a shared decision to initiate treatment, whichever comes first.
  Interventions: Other: Active Surveillance

INTERVENTIONS:
Other: Active Surveillance — Agreeing to postpone treatment while continuing with a CT scan surveillance regimen to follow tumor growth. SABR should be offered if either the tumor is >3 cm in size or the VDT decreases to <400 days.

SUMMARY:
Cancer patients are often given the choice of delaying or avoiding treatment as one of their options. However, there is not much information guiding lung cancer patients and their clinicians regarding this approach. Active surveillance is a way of either delaying or avoiding treatment and its possible side effects through carefully watching for changes in the tumor and considering treatment if there is progression. The purpose of this research study is to evaluate active surveillance and ways to better understand if and when to treat patients with stage IA lung cancer.

DETAILED DESCRIPTION:
The University of Vermont Medical Center is looking at determining if active surveillance is a viable option for low risk lung cancer patients. Currently, the National Cancer Care Network (NCCN) guidelines recommends considering stereotactic ablative radiotherapy (SABR) for patients not well enough for surgery, which is generally well tolerated, but it's also been shown to cause significant worsening of shortness of breath, fatigue, chest pain, and in extreme cases, death. Investigators are using this pilot study as a means to determine outcomes for patients who choose an active surveillance approach. This information could change future conversations between doctor and patient regarding treatment options, giving patients the choice to choose radiation therapy or to delay treatment by taking an active surveillance approach.

Investigators have published outcomes for 12 elderly patients with stage IA lung cancer who had chosen the active surveillance approach, reserving radiation therapy for when rapid tumor growth was determined (PMID 30648024). The clinical outcomes were similar to those expected if treatment had been provided, and at two years from the time the tumor was found almost half the patients were able to avoid getting radiation.

By deciding to participate in this study, patients are agreeing to postpone their treatment for an active surveillance approach while continuing with a computed tomography (CT) scan regimen to follow tumor growth. Once their tumor size is determined there are parameters in place to decide when patients should consider radiation. These parameters are based on speed of tumor growth over time and tumor size.

ELIGIBILITY:
Main Cohort Inclusion Criteria:

* Patient at UVMCC.
* Has pathologically proven recent diagnosis (≤180 days) of solitary or multifocal Stage T1a/b/c, N0, M0 [AJCC Staging, 8th Ed.] non-small cell lung cancer [NSCLC] or carcinoid tumors.
* History & physical ≤90 days prior to enrollment.
* Tumors may have a solid component of any magnitude ≤3 cm.
* Age ≥65 years old.
* Charlson Comorbidity Index [CCI] ≥6 within 90 days prior to enrollment.
* Zubrod performance status of 0-3 within 90 days prior to enrollment.
* Deemed unresectable or "medically inoperable" due to medical co-morbidities. Otherwise operable patients who decline surgery are considered inoperable.
* Eligible to receive treatment via SABR at the discretion of the treating oncologist.
* CT scan of the chest (contrast preferred) ≤90 days of enrollment with slice thickness ≤3 mm.
* Whole body PET scan ≤90 days prior to enrollment. [Preferably before biopsy performed]

Correlative Science Only Cohort Inclusion Criteria:

* Patient at UVMCC.
* Patients who have been followed via active surveillance > 180 days already may enroll in the correlative science only cohort for the purpose of blood draws only, regardless of reason active surveillance was chosen.
* Pathologically proven diagnosis (>180 days prior to enrollment) of solitary or multifocal Stage T1a/b/c, N0, M0 [AJCC Staging, 8th Ed.] non-small cell lung cancer [NSCLC] or carcinoid tumors.
* History & physical ≤90 days prior to enrollment.
* Any age.
* Any Charlson Comorbidity Index [CCI].
* Zubrod performance status of 0-3 within 90 days prior to enrollment.
* Can be medically operable or inoperable with any medical co-morbidities.
* CT scan of the chest (contrast preferred) ≤90 days around (before or after) enrollment with slice thickness ≤3 mm. [Frequency as deemed appropriate by managing oncologist].
* Whole body PET/CT scan [Not required pre-enrollment, and frequency as deemed appropriate by managing oncologist].

Exclusion Criteria (both cohorts):

* Prior radiation treatment of the study NSCLC.
* Prior receipt of any systemic treatment for the study NSCLC.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2018-07-31 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Primary Objective: Freedom-from radiation rate for patients on active surveillance | One year
  Freedom-from radiation rate for patients on active surveillance

SECONDARY OUTCOMES:
Secondary Objective: umber of participants on active surveillance with increased anxiety, depression, and uncertainty | Two years
  Number of participants on active surveillance with increased anxiety, depression, and uncertainty as assessed by the FACT-L, PROMIS-Fatigue, EQ-5D-5L, and State-Trait Anxiety Inventory questionnaires, change from baseline to end of study.

OTHER OUTCOMES:
Correlative Science Objective | Two years
  To correlate circulating tumor DNA [ctDNA], circulating tumor cells [CTCs], a cancer-associated macrophage-like cells [CAMLs] with disease aggressiveness as measured by VDT.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Vermont Medical Center, Burlington, Vermont, United States

REFERENCES:
- [Background] No HJ, Lester-Coll NH, Seward DJ, Sidiropoulos N, Gagne HM, Nelson CJ, Garrison GW, Kinsey CM, Lin SH, Anker CJ. Active Surveillance for Medically Inoperable Stage IA Lung Cancer in the Elderly. Cureus. 2018 Oct 22;10(10):e3472. doi: 10.7759/cureus.3472. PMID 30648024